CLINICAL TRIAL: NCT00641004
Title: Randomized Double-Blind Clinical Trial of Rebamipide vs Esomeprazole in the Treatment of NSAID-induced Gastropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Otsuka Pharmaceutical, Inc., Philippines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 037-PPB-0701i
Record Dates: First submitted 2008-03-18; First posted 2008-03-21 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2009-12

CONDITIONS: NSAID Induced Gastropathy
MeSH Terms: interventions — rebamipide; Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Rebamipide 100mg TID for 12 weeks
  Interventions: Drug: Rebamipide and Esomeprazole
- 2 (Active Comparator): Esomeprazole 40mg OD + Esomeprazole-matching placebo BID for 12 weeks
  Interventions: Drug: Rebamipide and Esomeprazole

INTERVENTIONS:
Drug: Rebamipide and Esomeprazole — 1. Rebamipide 100mg TID for 12 weeks
  2. Esomeprazole 40mg OD + Esomeprazole-matching placebo BID for 12 weeks

SUMMARY:
Primary objective: To determine the levels of malondialdehyde (MDA) and immunohistochemistry surrogate of inflammation in patients with NSAID-induced gastric mucosal injury treated with Rebamipide 3x a day vs Esomeprazole 40mg once a day. Secondary objective: For patients who become symptomatic during NSAID treatment, to compare the proportion of patients with positive treatment effects using the Likert scale. Third objective: To compare the proportion of patients with positive treatment effects as determined by Modified Lanza scoring between the two groups.

ELIGIBILITY:
Inclusion Criteria:

Patients with rheumatoid arthritis and osteoarthritis who developed dyspeptic symptoms while on NSAID for at leat 4 weeks who fulfill any of the following criteria: 1) Have not been on NSAIDs (NSAID-naïve) as they are newly diagnosed patients or satisfies ALL of the following criteria: a) Have not received NSAIDs for more than 2 years continuously, b) Have not received NSAID for at least 3 months, c) Does not take more than the therapeutic dose required for any of the following NSAIDS: Aspirin (at max. 4000mg.day), Naproxen (at max. 1375mg/day), Ibupropen (at max. 2400mg/day), Diclofenac (at max. 200mg/day), Piroxicam (at max. 40mg/day). 2) Gastric mucosal lesions on upper endoscopy (Lanza score ≥ 1) 3) More than 18 and less than 65 years old 4) Medically cleared and consents to undergo upper endoscopy 5) Willing to participate in the trial and sign an informed consent form

Exclusion Criteria:

1. Patients with known malignancy 2) Women who are pregnant and breastfeeding 3) Psychiatric illness 4) severe co-morbid illness like renal failure, cirrhosis, etc. 5) History of intake of any anti-secretory agent for the past 2 weeks 6) Patients with coagulation disorders and hematologic problems 7) Complicated ulcers, i.e. bleeding, perforating, etc. 8) Patients with evidence of portal hypertension i.e. varices, portal gastropathy, etc. 9) History of gastric surgery 10) Patients on COX-2 inhibitors 11) Modified Lanza score of 0 12) Herbal medications or complementary alternative medicines (e.g. glucosamine chondroitisulfate, etc. 13) (+)H.pylori test by RUT (Rapid Urease Test) and biopsy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine the levels of MDA and immunohistochemistry surrogate of inflammation in patients with NSAID-induced gastric mucosal injury. | Throughout the study

SECONDARY OUTCOMES:
For patients who become symptomatic during NSAID treatment, to compare the proportion of patients with positive treatment effects using the Likert scale | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Jose Sollano, MD, Principal Investigator — University of Santo Tomas Hospital
Locations (4):
- Philippines (4):
  - University of Santo Tomas Hospital, Manila
  - Armed Forces of the Philippines Medical Center, Quezon City
  - Veterans Memorial Medical Center, Quezon City
  - Candinal Santos medical Center, San Juan City